CLINICAL TRIAL: NCT01152905
Title: Effect of Nitrous Oxide on Cisatracurium Infusion Demands. A Randomized Controlled Trial.
Brief Title: Effect of Nitrous Oxide on Cisatracurium Infusion Demands
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Hanna Illman/Consultant Anesthesiologist, Dept. of Anaesthesiology, Intensive Care, Emergency Care and Pain Medicine
Other Study IDs: 225/2006
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2006-11

CONDITIONS: Neuromuscular Blocking Agents
Keywords: Neuromuscular blockade; Neuromuscular blocking agents; Atracurium; Nitrous oxide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Air/TIVA group: The patients received during the anesthesia a mixture of air with 30% oxygen All patients received total intravenous anesthesia (TIVA) using target controlled infusion of propofol and remifentanil.
- Nitrous oxide/TIVA group: The patients received nitrous oxide with 30% oxygen.All patients received total intravenous anesthesia (TIVA) using target controlled infusion of propofol and remifentanil.

SUMMARY:
Background: Recent studies have questioned our previous understanding on the effect of nitrous oxide on muscle relaxants, since nitrous oxide has been shown to potentiate the action of bolus doses of mivacurium, rocuronium and vecuronium. This study was aimed to investigate the possible effect of nitrous oxide on the infusion requirements of cisatracurium.

Methods: 70 ASA physical status I-III patients aged 18-75 years were enrolled in this randomized trial. The patients were undergoing elective surgery requiring general anesthesia with a duration of at least 90 minutes. Patients were randomized to receive propofol and remifentanil by target controlled infusion in combination with either a mixture of oxygen and nitrous oxide (Nitrous oxide/TIVA group) or oxygen in air (Air/TIVA group). A 0.1 mg/kg initial bolus of cisatracurium was administered before tracheal intubation, followed by a closed-loop computer controlled infusion of cisatracurium to produce and maintain a 90% neuromuscular block. Cumulative dose requirements of cisatracurium during the 90-min study period after bolus administration were measured and the asymptotic steady state rate of infusion to produce a constant 90% block was determined by applying nonlinear curve fitting to the data on the cumulative dose requirement during the study period.

Results: Controller performance, i.e. the ability of the controller to maintain neuromuscular block constant at the setpoint and patient characteristics were similar in both groups. The administration of nitrous oxide did not affect cisatracurium infusion requirements. The mean steady-state rates of infusion were 0.072 +/- 0.018 and 0.066 +/- 0.017 mg * kg-1 * h-1 in Air/TIVA and Nitrous oxide/TIVA groups, respectively.

Conclusions: Nitrous oxide does not affect the infusion requirements of cisatracurium.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III patients

Exclusion Criteria:

* Patients with significant renal,
* Hepatic or cardiac disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery requiring general anesthesia with a duration of at least 90 minutes.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2007-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Intensive Care, Emergency Care and Pain Medicine, Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Illman HL, Antila HM, Olkkola KT. Effect of nitrous oxide on cisatracurium infusion demands: a randomized controlled trial. BMC Anesthesiol. 2010 Aug 18;10:14. doi: 10.1186/1471-2253-10-14. PMID 20718983